CLINICAL TRIAL: NCT02797002
Title: Validity of Neck Extensor Muscles Endurance Test in Non-specific Chronic Neck Pain and Asymptomatic Subjects
Status: Completed | Type: Observational
Sponsor: University of Social Welfare and Rehabilitation Science (Other)
Responsible Party: Principal Investigator, Dr. L. Ghamkhar, PhD Candidate, University of Social Welfare and Rehabilitation Science
Other Study IDs: IR.USWR.REC.1394.191
Record Dates: First submitted 2016-06-03; First posted 2016-06-13 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Chronic non specific neck pain: Experiencing neck pain for at least 3 months in the last year
  Interventions: Other: Assessment
- Without neck pain (asymptomatic): No history of neck pain
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment

SUMMARY:
Neck pain (NP) is one of the most common and costly musculoskeletal complaints in today's societies. Cervical muscles endurance has been commonly associated with the development of NP. Real-time ultrasound imaging is a reliable and valid technique recently used by physical therapists to evaluate muscle structure, function and activation patterns. The aim of this study is if change in muscle thickness can correlate with the results of the endurance testing.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with neck pain: experiencing pain for at least 3 months in the last year, having pain score of 3 or more on visual analogue scale.
* Healthy subjects: no history of neck pain

Exclusion Criteria:

* History of cervical discopathy
* Any surgery on neck
* Traumatic neck injury
* Any congenital disorders

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects with and without neck pain
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2015-03; Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Flexor and Extensor cervical muscles holding time (second) | 6 months
Anteroposterior diameter of the flexor and extensor cervical muscles (mm) | 6 months
Mediolateral diameter of the flexor and extensor cervical muscles (mm) | 6 months
Cross section area of the flexor and extensor cervical muscles (cm2) | 6 months
Neck disability questionnaire score | 6 months
Visual analogue scale score | 6 months

SECONDARY OUTCOMES:
Pearson correlation coefficient of the cervical muscles holding time with Anteroposterior and border and cross section area of the flexor and extensor cervical muscles | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Social Welfare and Rehabilitation Sciences, Tehran, Iran